CLINICAL TRIAL: NCT02558023
Title: The Treatment of Hypertension Associated With Severe Preeclampsia. A Randomize Controlled Trial of Urapidil Versus Nicardipine. The Uranic Trial
Brief Title: The Treatment of Hypertension Associated With Severe Preeclampsia (PE). A Trial of Urapidil Versus Nicardipine
Acronym: Uranic
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: no candidats
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5866
Record Dates: First submitted 2015-08-24; First posted 2015-09-23 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2019-08

CONDITIONS: Hypertension; Preeclampsia
Keywords: PRE-ECLAMPSIA; URAPIDIL; NICARDIPINE
MeSH Terms: conditions — Hypertension; Pre-Eclampsia | interventions — urapidil; Nicardipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urapidil (Experimental): Urapidil (Eupressyl*) : IV One initial iv bolus of 12.5 mg. One or more bolus of 6.25 mg at intervals of 5 minutes if the diastolic pressure remains above 100 mmHg.
  The treatment is then continued at 4 mg.h-1 iv via a syringe pump. The maintenance dose needed to maintain MAP between 100 and 120 mmHg is sought by adjustments of ± 2 mg.h-1every 5 minutes.
  Maximum dose of 30 mg.h-1.
  Interventions: Drug: Urapidil
- Nicardipine (Active Comparator): Nicardipine : IV
  1 mcg.kg-1.min-1until reduction MAP 15%. Reduction 1/4 of the posology (0.75 mcg.kg -1.min-1). The maintenance dose needed to maintain MAP between 100 and 120 mmHg is then sought by adjustments of ± 0.25 mcg.kg.min-1every 5 minutes.
  Maximum dose of 6 mg.h-1
  Interventions: Drug: Nicardipine

INTERVENTIONS:
Drug: Urapidil — Urapidil (Eupressyl*) : IV One initial iv bolus of 12.5 mg. One or more bolus of 6.25 mg at intervals of 5 minutes if the diastolic pressure remains above 100 mmHg.
  The treatment is then continued at 4 mg.h-1 iv via a syringe pump. The maintenance dose needed to maintain MAP between 100 and 120 mmHg is sought by adjustments of ± 2 mg.h-1every 5 minutes.
  Maximum dose of 30 mg.h-1.
  Arms: Urapidil
Drug: Nicardipine — Nicardipine : IV
  1 mcg.kg-1.min-1until reduction MAP 15%. Reduction 1/4 of the posology (0.75 mcg.kg -1.min-1). The maintenance dose needed to maintain MAP between 100 and 120 mmHg is then sought by adjustments of ± 0.25 mcg.kg.min-1every 5 minutes.
  Maximum dose of 6 mg.h-1
  Arms: Nicardipine

SUMMARY:
The objective of this study is to demonstrate that urapidil is not inferior to nicardipine for the treatment of hypertension associated with preeclampsia (PE) and that it is better tolerated.

* efficacy endpoint : mean arterial blood pressure corrected to 100-120 mmHg after 120 min of study drug administration.
* safety endpoints : clinical and biological observation for any side effect. All infants will be observed in the neonatology unit (during 48h).

Pharmacokinetic study included to study :

* transplacental transfer,
* transfer in breast milk,
* and neonatal elimination (premature babies of mothers treated with urapidil (less than 33 WG))

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Singleton pregnancy
* Patients with remaining hypertension despite an oral treatment for who an iv antihypertensive treatment is indicated

Patient with PE, as defined by :

* Systolic Blood Pressure (BP) ≥ 140 mmHg and/or Diastolic BP ≥ 90 mmHg, after the 20th week of amenorrhea, without chronic hypertension, AND
* Proteinuria > 300 mg.day-1 or > 2 crosses(++) on an urinary dipstick,

OR

Patient with severe Pregnancy Induced Hypertension (PIH), as defined by :

Systolic BP ≥ 160 mmHg and/or Diastolic BP ≥110 mmHg, after the 20th week of amenorrhea, without chronic hypertension,

* Written informed consent signed and dated by both investigator and patient,
* Valid social security affiliation

Exclusion Criteria:

* Known allergy to study drugs
* Contra-indication to the study drugs: stenosis of the aortic isthmus, arteriovenous shunt, coarctation of the aorta, unstable angina, compensatory hypertension, myocardial infarction < 8 days.
* Eclampsia
* Person with difficulty understanding information
* Person with diminished responsibility,
* Ongoing intravenous antihypertensive treatment,
* No pressure cuff adapted to the morphology of the arms of the patients
* Concomitant use of 5 phosphodiesterase inhibitors
* Participation in a clinical trial within 6 months prior to inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Blood pressure at two hours | up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DIEMUNSCH, PUPH, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service d'Anesthésie - CMCO, Schiltigheim
  - Service d'Anesthésie et de Réanimation Médicale, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg